CLINICAL TRIAL: NCT06073028
Title: Model-based Cueing-as-needed for Walking in Parkinson's Disease
Acronym: GAITPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Emilie Hutin, Director, Henri Mondor University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GAITPARK
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Walking, Difficulty; Gait, Festinating
Keywords: Basal Ganglia Diseases; Gait analysis; Gait Speed; Cues; Exercise Therapy
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation; Gait Disorders, Neurologic; Basal Ganglia Diseases

STUDY DESIGN:
Intervention Model Description: Pilot single-blind randomized cross-over study, with the subject blind as to the hypothesis
Who Masked: Outcomes Assessor
Masking Description: A biomechanics engineer leads the gait assessment, being blinded to the allocation schedule, and participants were specifically asked to not discuss the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic auditory cueing (Experimental): The rhythmic auditory cueing (RAC) is a constant stimulation ("bip" signal) delivered by a numeric metronome, which is adjusted on 110% of the patient's own cadence.
  Interventions: Other: 20-minute gait training
- Adaptive spatial auditory cueing (Experimental): Adaptive spatial auditory cueing (ASAC) is a verbal instruction stimulation delivered by an application when the stride length of the patient is less than a predetermined threshold, during two consecutive strides. The instruction is given in the patient's native language, which is French: "allongez le pas" (i.e. "lengthen the step"). The predetermined threshold is 110% of the patient's own stride length.
  Interventions: Other: 20-minute gait training

INTERVENTIONS:
Other: 20-minute gait training — All subjects undergo two 20-minute gait trainings using two different kinds of auditory cueing (temporal or spatial), one week apart (D1 and D8).

SUMMARY:
Correcting of the lack of regularity in steps is a key component of gait rehabilitation in Parkinson's disease. The proposal is to introduce adaptive spatial auditory cueing (ASAC) based on verbal instruction "lengthen the step" automatically delivered when the stride length decreased below a predetermined threshold. The present study compared the effect of usual rhythmic auditory cueing versus ASAC used during a walking training in Parkinson's disease.

DETAILED DESCRIPTION:
Correcting of the lack of regularity in steps is a key component of gait rehabilitation in Parkinson's disease. The proposal is to introduce adaptive spatial auditory cueing (ASAC) based on verbal instruction "lengthen the step" automatically delivered when the stride length decreased below a predetermined threshold. The present study compared the effect of usual rhythmic auditory cueing versus ASAC used during a walking training in Parkinson's disease. Fifteen patients with Parkinson's disease performed both interventions in randomized order, one week apart: a 20-minute walking training with rhythmic auditory cueing, in form of a metronome adjusted on 110% of the patient's own cadence, or ASAC delivered when the stride length is less than 110% of the patient's own stride length. Assessment criteria were walking distance covered during the intervention, speed, step length, cadence, coefficients of variation of step length and step duration, and indexes of spatial and temporal asymmetry during a walking test before and just after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of idiopathic PD based on the United Kingdom-Parkinson's Disease Society Brain Bank criteria;
* stage 2 or 3 on the Hoehn and Yahr scale;
* comfortable walking speed over 10 meters ≤ 1 m/s;
* ability to walk over 20 minutes without aids or antiparkinsonian medications;
* a stable antiparkinsonian medication regime;
* cognitive abilities to understand the verbal instructions for a walking test according to the investigator's judgment;
* written consent for the participation.

Exclusion Criteria:

* intercurrent disease other than PD, affecting gait;
* any intercurrent medical condition preventing them from participating in two consecutive gait training one week apart;
* medical diagnosis of hearing loss;
* non-affiliation to the social security regime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Walking speed | Before and just after the intervention
  Speed in free walking condition over 10 meters barefoot, without any assistance

CONTACTS AND LOCATIONS:
Overall Officials: Hutin Emilie, PhD, Principal Investigator — HenriMondorHU
Locations (1):
- Laboratoire Analyse et Restauration du Mouvement, Créteil, France

IPD SHARING:
Plan to Share IPD: No